CLINICAL TRIAL: NCT06092957
Title: Reduced-dose Radiotherapy With/Without Concurrent Chemotherapy Versus Standard Chemoradiotherapy for High-risk Locoregionally Advanced Nasopharyngeal Carcinoma Who Achieved Complete Response After Induction Chemotherapy Plus Immunotherapy: a Randomized, Open-label, Multicenter, Phase III Trial
Brief Title: Reduced-dose RT With/Without CCT Versus Standard CCRT for High-risk LANPC Who Achieved CR Post Induction Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Guangdong Provincial People's Hospital (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); The fifth Affiliated Hospital of Guangzhou Medcial University (Other Government); Zhongshan People's Hospital, Guangdong, China (Other); Hunan Cancer Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2023-09-25
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Nasopharyngeal Carcinoma; De-escalation Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Induction chemotherapy plus conventional concurrent chemoradiotherapy (Active Comparator)
  Interventions: Drug: Cisplatin-based induction chemotherapy; Drug: Full course of PD-1/PD-L1 blockades; Radiation: Standard-dose IMRT; Drug: Concurrent Chemotherapy
- Induction chemotherapy plus reduced-dose radiotherapy and concurrent chemotherapy (Experimental)
  Interventions: Drug: Cisplatin-based induction chemotherapy; Drug: Full course of PD-1/PD-L1 blockades; Radiation: Reduced-dose IMRT; Drug: Concurrent Chemotherapy
- Induction chemotherapy plus reduced-dose radiotherapy alone (Experimental)
  Interventions: Drug: Cisplatin-based induction chemotherapy; Drug: Full course of PD-1/PD-L1 blockades; Radiation: Reduced-dose IMRT

INTERVENTIONS:
Drug: Cisplatin-based induction chemotherapy — Cisplatin-based induction chemotherapy will be given every 3 weeks for 3 cycles before radiotherapy including GP, TP, and TPF regimen.
Drug: Full course of PD-1/PD-L1 blockades — a) Camrelizumab 200mg, b) Toripalimab 240mg, or c) Adebrelimab 1200mg will be started on day 1 of induction chemotherapy and given every 3 weeks for up to 12 cycles, or until intolerable toxicity, or disease progression or withdrawal from the treatment.
Radiation: Reduced-dose IMRT — GTVnx:60Gy/30F/2.0Gy，CTV1:54Gy/30F/1.8Gy，CTV2:48Gy/30F/1.6Gy
  Arms: Induction chemotherapy plus reduced-dose radiotherapy alone; Induction chemotherapy plus reduced-dose radiotherapy and concurrent chemotherapy
Radiation: Standard-dose IMRT — GTVnx：69.96Gy/33Fr/2.12Gy；CTV1：60.60Gy/33Fr/1.82y；CTV2：54.12Gy/33Fr/1.64Gy
  Arms: Induction chemotherapy plus conventional concurrent chemoradiotherapy
Drug: Concurrent Chemotherapy — Cisplatin 100mg/m2 every 3 weeks for 2 cycles
  Arms: Induction chemotherapy plus conventional concurrent chemoradiotherapy; Induction chemotherapy plus reduced-dose radiotherapy and concurrent chemotherapy

SUMMARY:
This prospective trial aims to enroll patients with high-risk stage III-IVA (AJCC 8th, except T3N0) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Under the condition of full course of PD-1/PD-L1 blockades, patients who achieved both radiological and biological complete response after 3 cycles of platinum-based chemotherapy plus PD-1/PD-L1 blockades will be randomized in a 1:1:1 ratio to receive reduced-dose radiotherapy (60Gy/30F) alone or reduced-dose radiotherapy plus concurrent chemotherapy or standard dose radiotherapy (70Gy/33F) with concurrent chemotherapy. To solve the urgent problem of whether patients with high-risk advanced nasopharyngeal carcinoma are suitable for downgrade treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
2. Tumor staged as III-IVA (AJCC 8th, except T3N0).
3. Patients who achieved both radiological and biological CR according to the RECIST criteria on the basis of MRI, PET-CT and endoscopic biopsy, and EBV DNA load =0 copies/mL (or lower than the test line) after 3 cycles of induction therapy of platinum-based chemotherapy plus immunotherapy.
4. Eastern Cooperative Oncology Group performance status ≤1.
5. Adequate organ function:

   Adequate marrow function: neutrocyte count≥4×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.

   Adequate liver and kidney function: Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 2.5×ULN.; creatinine clearance rate ≥ 60 ml/min or creatinine of no more than 1.5 times the upper normal limit.
6. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients who are evaluated as PR or SD or PD or EBV DNA load of >0 copies/mL after 3 cycles of induction therapy of platinum-based chemotherapy plus PD-1/PD-L1 blockades.
2. The laboratory examination value does not meet the relevant standards within 7 days before enrollment.
3. Patients have received prior chemotherapy, immunotherapy, targeted therapy, or surgery (other than diagnostic treatment).
4. Subjects who underwent anti-PD-1 /PD-L1 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell synergistic stimulation or checkpoint pathway) and anti-angiogenic drugs.
5. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease).
6. Grade ≥2 epistaxis (defined as the need for medical intervention such as nasal tamponade, cautery, topical vasoconstrictors, according to CTCAE 5.0) within 1 month prior to enrollment; Macroscopic hemoptysis or hematemesis) is defined as ≥1/2 teaspoon of bright red blood, or a blood clot with little/no sputum on each cough). (Patients with mixed sputum-blood occasionally may be enrolled).
7. Patients with hypertension who cannot be reduced to the normal range by antihypertensive drug treatment (systolic blood pressure > 140 mmHg/diastolic blood pressure > 90 mmHg), patients with ≥ grade II coronary heart disease, arrhythmia (including QTc interval prolongation > 450 ms in men and > 470 ms in women) and cardiac insufficiency.
8. Patients currently take warfarin, heparin, aspirin (> 325 mg/day) or other NSAIDs known to inhibit platelet function, ticlopidine, clopidogrel, or cilostazol. (Patients can be enrolled if they discontinue these drugs 10 days prior to the commence of study and meet the requirements of coagulation in the enrollment criteria).
9. Patients with other malignancies (except for cervical cancer, basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer, and ductal carcinoma in situ who have undergone curative treatment).
10. Has a known history of interstitial lung disease.
11. Known history of hypersensitivity to any components of the PD-1/PD-L1 blockades formulation or other monoclonal antibodies.
12. Has a known history of allergic reactions to the drugs in the study (gemcitabine, cisplatin, docetaxel, abraxane, paclitaxel ).
13. Has active autoimmune disease or any condition that requires systemic corticosteroid or immunosuppressive therapy, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval.
14. Complications requiring long-term use of immunosuppressive drugs or systemic or local use of immunosuppressive-dose corticosteroids.
15. HIV positive; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C with blood screening positive (HCV antibody positive).
16. Has a known history of active TB (bacillus tuberculosis) within 1 year; anti-TB treatment is ongoing or within 1 year prior to screening.
17. Has received a live vaccine; or a systematic glucocorticoid therapy ; or any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) ; any Chinese anti-tumor herbs within 4 weeks prior to enrollment.
18. Pregnancy or breastfeeding.
19. Other patients who were considered unsuitable by the treating physicians.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
The proportion of patients with treatment related acute complications | 1 year
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
The proportion of patients with treatment related late complications | 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China